CLINICAL TRIAL: NCT00748202
Title: Pharmacokinetics Berinert P Study of Subcutaneous Versus Intravenous Administration in Subjects With Moderate Hereditary Angioedema - The Passion Study
Brief Title: Berinert P Study of Subcutaneous Versus Intravenous Administration
Acronym: PASSION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Clinical trial center Rhine-Main (Unknown); ZKI Kindergerinnungslabor (Other); Institut für Medizinische Virologie JWG-University hospital (Unknown); CSL Behring (Industry); PharmaPart (Industry); University of Milan (Other)
Responsible Party: PD Dr. Wolfhart Kreuz, Centre of Paediatrics III, Department of Haematology, Haemostaseology and Oncology, Comprehensive Care Centre for Thrombosis and Haemostasis
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CE1145_1001
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; C1-Esterase inhibitor; intravenous; subcutaneous; pharmacokinetic
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): intravenous administration of C1-Inhibitor, after the end of the first observation period (at least after 7 days), each arm switches cross-over to the alternative administration mode not investigated so far
  Interventions: Drug: C1-Esterase Inhibitor
- 2 (Active Comparator): subcutaneous administration of C1-Inhibitor. After the end of the first observation period (at least after 7 days), each arm switches cross-over to the alternative administration mode not investigated so far.
  Interventions: Drug: C1-Esterase Inhibitor

INTERVENTIONS:
Drug: C1-Esterase Inhibitor — 1000 I.E.
  Other Names: Berinert P

SUMMARY:
The study is performed to investigate the subcutaneous (s.c.) versus intravenous (i.v.) administration of Berinert P in patients with hereditary angioedema (HAE) to establish a second administration mode in cases where i.v. access is not suitable.

The study is planned as a single centre, randomized, open-label, cross-over pharmacokinetic study.

Subjects will either start with s.c. or i.v. pasteurised C1-Inhibitor concentrate (Berinert P) and than switch to the treatment not administered before.

DETAILED DESCRIPTION:
Patients with hereditary angioedema (HAE), suffer from recurring and mostly unforeseeable attacks of acute oedema of subcutaneous tissues of various organs. The pathophysiological correlate of this disease is a deficiency in functionally active C1-Esterase Inhibitor (C1-INH). Today, two main types of HAE are described. In HAE type I, an impaired synthesis and an elevated turnover of a normal and functional active C1-INH molecule takes place, causing reduced amounts in functionally active C1-INH. In HAE type II, normal levels of a functionally impaired C1-INH molecule are synthesized. Both defects are inherited as an autosomal dominant trait. HAE type III is limited to females and not associated with C1-INH deficiency; the pathophysiology of this type remains to be determined. Corticosteroids, antihistamines or epinephrine usually do not exert any positive effect in acute attacks caused by HAE. This is of particular importance as these types of medication are often used in case of oedema in general. In case of acute oedema in patients suffering from HAE, the intravenous administration of C1-INH concentrate (e.g., Berinert P) is the treatment of choice. The study is performed to investigate the s.c. versus i.v. administration of Berinert P in patients with hereditary angioedema (HAE) to establish a second administration mode in cases where i.v. access is not suitable.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an established diagnosis of HAE type I (C1-Inhibitor activity < 50% and C1-Inhibitor antigen < 15.4 mg/dl) or HAE type II (C1-Inhibitor activity < 50% and C1-Inhibitor antigen in normal or elevated concentration of dysfunctional protein).
* Male and female subjects with an age of at least 18 years.
* Subjects providing an informed consent.

Exclusion Criteria:

* Subjects without an established diagnosis of HAE.
* Last C1-INH administration less than 7 days ago and/or acute attack.
* Subjects with acquired angioedema (AAE).
* All other types of angioedema not associated with C1-INH deficiency.
* Treatment with any investigational drug (exclusive drugs appropriate for the treatment of acute angioedema) 30 days before study treatment.
* Treatment with any other drug appropriate for the treatment of acute angioedema within 7 days before start of study treatment at each phase.
* Danazol prophylaxis.
* Prophylaxis with antifibrinolytics, EACA, tranexamic acid.
* Subjects with a known hypersensitivity to study medication (Berinert P).
* Pregnant women (pregnancy rapid assay required for women with childbearing potential), women currently breast-feeding, or with the intention to breast-feed
* Subjects with malignant diseases.
* Subjects with immunodeficiencies such as established acquired immunodeficiency syndrome.
* Subjects with concurrent serious or acute illness or infection as per investigators judgement.
* Subjects with mental conditions which render the subject or its legally acceptable representative unable to understand the nature, scope and possible consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Individual courses of C1-inhibitor levels, from these will be derived pharmacokinetic parameters | i.v. and s.c.samples: 0, 0.25, 0.5, 0.75 hours and 1, 2, 4, 6, 8, 12, 16, 20, 24, 36, 48, 60, 72, 120, 168, 336 an 504 hours.

SECONDARY OUTCOMES:
Safety of s.c. and i.v. administration of study medication | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wolfhart Kreuz, PD Phd, Principal Investigator — Centre of Paediatrics III, Department of Haematology, Haemostaseology and Oncology, Comprehensive Care Centre for Thrombosis and Haemostasis, Johann-Wolfgang-Goethe-University Hospital
Locations (1):
- Centre of Paediatrics III, Department of Haematology, Haemostaseology and Oncology, Comprehensive Care Centre for Thrombosis and Haemostasis, Johann-Wolfgang-Goethe-University Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Martinez-Saguer I, Cicardi M, Suffritti C, Rusicke E, Aygoren-Pursun E, Stoll H, Rossmanith T, Feussner A, Kalina U, Kreuz W. Pharmacokinetics of plasma-derived C1-esterase inhibitor after subcutaneous versus intravenous administration in subjects with mild or moderate hereditary angioedema: the PASSION study. Transfusion. 2014 Jun;54(6):1552-61. doi: 10.1111/trf.12501. Epub 2013 Nov 24. PMID 24266596